CLINICAL TRIAL: NCT05031338
Title: Carpal Tunnel Release Using Ultrasound Patient Experience Registry
Brief Title: Carpal Tunnel Release Using Ultrasound
Acronym: CiTRUS
Status: Terminated | Type: Observational
Why Stopped: Sponsor changing database systems for ease of use for patient data collection
Sponsor: Sonex Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL002
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Release; Ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SX-One MicroKnife with ultrasound guidance: Carpal Tunnel Release using the SX-One MicroKnife with ultrasound guidance
  Interventions: Device: Carpal Tunnel Release; Procedure: Carpal Tunnel Release
- Traditional mini-open technique without ultrasound guidance: Carpal Tunnel Release using the traditional mini-open technique without ultrasound guidance
  Interventions: Device: Carpal Tunnel Release; Procedure: Carpal Tunnel Release

INTERVENTIONS:
Device: Carpal Tunnel Release — Carpal Tunnel Release surgery involves transecting the transverse carpal ligament (TCL) in order to reduce median nerve compression and alleviate symptoms. The carpal tunnel release surgery will be performed using the SX-One MicroKnife with ultrasound guidance.
Procedure: Carpal Tunnel Release — Carpal Tunnel Release surgery involves transecting the transverse carpal ligament (TCL) in order to reduce median nerve compression and alleviate symptoms. The carpal tunnel release surgery will be performed using the traditional mini-open technique without ultrasound guidance.

SUMMARY:
The goal of the Carpal Tunnel Release Using Ultrasound registry (CiTRUS Registry) is to collect experience information from patients scheduled to undergo carpal tunnel release surgery with either the SX-One MicroKnife® with ultrasound guidance or the traditional mini-open technique without US guidance.

DETAILED DESCRIPTION:
The CiTRUS registry is an observational study designed to better understand the overall patient experience following a carpal tunnel release surgery using either the SX-One MicroKnife with ultrasound guidance or the traditional mini-open technique without ultrasound guidance. The determination of which surgical technique to uses will be determined by the treating physician and the patient. The patient registry outcomes are intended to help direct future clinical care, educate patients with carpal tunnel syndrome, and design future research.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo carpal tunnel release surgery on the right and/or left wrist using either the SX-One MicroKnife with US guidance or the traditional mini-open technique without US guidance
* 18 years of age or older
* Agree to complete questionnaires over a 12-month period
* Valid mobile phone number and email address to receive and answer questions

Exclusion Criteria:

• Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo carpal tunnel release surgery using either the SX-One MicroKnife® with ultrasound (US) guidance or the traditional mini-open technique without ultrasound guidance.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Quick Form of the Disabilities of the Shoulder and Hand scores at 12 months | 12 months
  To assess the overall patient experience following carpal tunnel release using either the SX-One MicroKnife® with ultrasound (US) guidance or the traditional mini-open technique without ultrasound guidance patients will complete the Quick Form of the Disabilities of the Shoulder and Hand scale. The Quick Form of the Disabilities of the Shoulder and Hand scale consists of 11 items scored 1-5 with lower scores indicating less symptoms or better function.
Change from baseline Boston Carpal Tunnel Questionnaire scores at 12 months | 12 months
  To assess the overall patient experience following carpal tunnel release using either the SX-One MicroKnife® with ultrasound guidance or the traditional mini-open technique without ultrasound guidance patients will complete the Boston Carpal Tunnel Questionnaire at 12 months. The Boston Carpal Tunnel Questionnaire consists of two subscales: symptom severity (11 items scored 1-5) and functional status (8 items scored 1-5) with lower scores indicating less symptoms or better function.

SECONDARY OUTCOMES:
Patient reported time to return to activities | Post-operative days 1-14, 2 weeks, 1,3,6 and 12 months
  Patient reported time to return to normal activities as measured in days.

OTHER OUTCOMES:
Patient reported satisfaction following carpal tunnel release | 2 weeks, 1,3,6 and 12 months
  Patient reported satisfaction with the carpal tunnel release procedure on a 1-5 scale with higher numbers indicating greater satisfaction.
Patient reported symptom improvement following carpal tunnel release | 2 weeks, 1,3,6 and 12 months
  Patient reported improvement in symptoms following carpal tunnel release, reported on a 1-5 scale with higher numbers indicating more symptom improvement.
Pain reported pain on numerical pain rating scale | Post-operative days 1-14, 2 weeks, 1,3,6 and 12 months
  Patient reported pain following carpal tunnel release, reported on an 11-point (0-10) numerical pain rating scale with higher numbers indicating more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Smith, MD, Principal Investigator — Sonex Health, Inc.
Locations (1):
- Sonex Health, Inc., Eagan, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamel SI, Freid B, Pomeranz C, Halpern EJ, Nazarian LN. Minimally Invasive Ultrasound-Guided Carpal Tunnel Release Improves Long-Term Clinical Outcomes in Carpal Tunnel Syndrome. AJR Am J Roentgenol. 2021 Aug;217(2):460-468. doi: 10.2214/AJR.20.24383. Epub 2020 Sep 2. PMID 32876476
- [Background] Chappell CD, Beckman JP, Baird BC, Takke AV. Ultrasound (US) Changes in the Median Nerve Cross-Sectional Area After Microinvasive US-Guided Carpal Tunnel Release. J Ultrasound Med. 2020 Apr;39(4):693-702. doi: 10.1002/jum.15146. Epub 2019 Oct 29. PMID 31659789
- [Background] Joseph AE, Leiby BM, Beckman JP. Clinical Results of Ultrasound-Guided Carpal Tunnel Release Performed by a Primary Care Sports Medicine Physician. J Ultrasound Med. 2020 Mar;39(3):441-452. doi: 10.1002/jum.15120. Epub 2019 Aug 26. PMID 31449326
- [Background] Henning PT, Yang L, Awan T, Lueders D, Pourcho AM. Minimally Invasive Ultrasound-Guided Carpal Tunnel Release: Preliminary Clinical Results. J Ultrasound Med. 2018 Nov;37(11):2699-2706. doi: 10.1002/jum.14618. Epub 2018 Apr 2. PMID 29608024
- [Background] Latzka EW, Henning PT, Pourcho AM. Sonographic Changes After Ultrasound-Guided Release of the Transverse Carpal Ligament: A Case Report. PM R. 2018 Oct;10(10):1125-1129. doi: 10.1016/j.pmrj.2018.02.018. Epub 2018 Mar 6. PMID 29518589
- [Background] Henning T, Lueders D, Chang K, Yang L. Ultrasound-Guided Carpal Tunnel Release Using Dynamic Expansion of the Transverse Safe Zone in a Patient With Postpolio Syndrome: A Case Report. PM R. 2018 Oct;10(10):1115-1118. doi: 10.1016/j.pmrj.2018.02.016. Epub 2018 Mar 6. PMID 29518587
- [Background] Leiby BM, Beckman JP, Joseph AE. Long-term Clinical Results of Carpal Tunnel Release Using Ultrasound Guidance. Hand (N Y). 2022 Nov;17(6):1074-1081. doi: 10.1177/1558944720988080. Epub 2021 Jan 29. PMID 33511873